CLINICAL TRIAL: NCT02869815
Title: Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy Using the Navigation of the Combination of Indocyanine and Blue Dye in Patients With Breast Cancer
Brief Title: ICG and Blue Dye Guided Sentinel Lymph Node Biopsy in Patients Underwent Neoadjuvant Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKUPHSLN003
Record Dates: First submitted 2016-07-29; First posted 2016-08-17 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Breast Neoplasms
Keywords: Methylene blue; Indocyanine green; Neoadjuvant Therapy; Sentinel Lymph Node Biopsy; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICG+Methylene Blue: ICG+Methylene Blue:
  Sentinel Lymph Node (SLN) identification and resection using dual tracer technique with the sub-areolar injection of ICG+Blue dye, before surgery.
  Interventions: Procedure: ICG+Methylene Blue

INTERVENTIONS:
Procedure: ICG+Methylene Blue — ICG+Methylene Blue Arm:
  One ml of methylene blue (1%) would be in injected sub-areolarly 5 minutes before surgery, and 1ml of ICG (0.125%) in the same site 3 minutes later. Massage of the breast would be applied to facilitate the movement of the tracers. A small incision would be made in the axilla, and a special device would be used to search the light nodes. During the sampling, blue nodes would also be resected . After the completion of SLNB, complete axillary dissection would be carried out.

SUMMARY:
The value of sentinel lymph node biopsy (SLNB) in patients underwent neoadjuvant chemotherapy is controversial. Lower detection rate and higher false negative rate are the main problem. The purpose of this study is to determine the detection rate and the false negative rate of SLNB by indocyanine green (ICG) in addition to blue dye (methylene blue) after neoadjuvant chemotherapy in patients with large or locally advanced breast cancer. This is a single arm clinical trial.

DETAILED DESCRIPTION:
Patients indicated for neoadjuvant therapy would be recruited in this study. During the surgery, SLNB using the dual tracing method would be applied before axillary clearance. After the surgery, histological results of the SLN and non-SLN would be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for neoadjuvant therapy
* Have complete evaluation of the axillary status
* Planned for axillary clearance after neoadjuvant therapy

Exclusion Criteria:

* Sensitive to Iodine
* Inflammatory disease
* Patient's refusal to join the trial

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with large operable or locally advanced breast cancer underwent neoadjuvant therapy.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Detection rate of SLN | Immediate
  The number of successful SLNB / total number of SLNB

SECONDARY OUTCOMES:
False negative rate of SLNB | 1 week after the surgery
  The number of patients with positive SLN / the number of patients with positive node
Adverse effect | Half a year after the surgery
  Prophylaxis reaction, skin complication

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Breast Center, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuehn T, Bauerfeind I, Fehm T, Fleige B, Hausschild M, Helms G, Lebeau A, Liedtke C, von Minckwitz G, Nekljudova V, Schmatloch S, Schrenk P, Staebler A, Untch M. Sentinel-lymph-node biopsy in patients with breast cancer before and after neoadjuvant chemotherapy (SENTINA): a prospective, multicentre cohort study. Lancet Oncol. 2013 Jun;14(7):609-18. doi: 10.1016/S1470-2045(13)70166-9. Epub 2013 May 15. PMID 23683750
- [Background] Boughey JC, Suman VJ, Mittendorf EA, Ahrendt GM, Wilke LG, Taback B, Leitch AM, Kuerer HM, Bowling M, Flippo-Morton TS, Byrd DR, Ollila DW, Julian TB, McLaughlin SA, McCall L, Symmans WF, Le-Petross HT, Haffty BG, Buchholz TA, Nelson H, Hunt KK; Alliance for Clinical Trials in Oncology. Sentinel lymph node surgery after neoadjuvant chemotherapy in patients with node-positive breast cancer: the ACOSOG Z1071 (Alliance) clinical trial. JAMA. 2013 Oct 9;310(14):1455-61. doi: 10.1001/jama.2013.278932. PMID 24101169
- [Derived] Liu M, Yang Y, Hua B, Feng R, Xu T, Wang M, Qi X, Cao Y, Zhou B, Tong F, Liu P, Liu H, Cheng L, Yang H, Xie F, Wang S, Wang C, Peng Y, Shen D, Chen L, Jiang J, Wang S. Indocyanine Green Fluorescence Plus Blue Dye for Sentinel Lymph Node Biopsy in Patients Undergoing Neoadjuvant Chemotherapy for Breast Cancer: A Multicenter, Prospective Cohort Study. Thorac Cancer. 2025 Jan;16(2):e15511. doi: 10.1111/1759-7714.15511. Epub 2024 Dec 27. PMID 39731298